CLINICAL TRIAL: NCT01218035
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy of Zoledronic Acid in Enhancement of Early Stability of Cementless Primary Hip Prosthesis
Brief Title: Efficacy of Zoledronic Acid in Enhancement of Early Stability of Cementless Primary Hip Prosthesis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Academy of Finland (Other); Novartis (Industry); Stryker Nordic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 94/180/2006
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Hip Osteoarthritis
Keywords: Hip osteoarthritis; Bisphophonate therapy; Zoledronic acid; Radiostereometric analysis; Osteoporosis
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoporosis | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: zoledronic acid — The patients in the active-treatment group will receive a single 5 mg dose of zoledronic acid intravenously just prior to release from the hospital (about 5th day post-surgery) as an adjunct therapy. The control group will receive a placebo (saline) infusion. All infusions will be given 100 ml in volume and infused over a period of 15 minutes with a pre- and post-infusion flush with normal saline.

SUMMARY:
This is a randomized, double-blind and placebo-controlled study to evaluate the efficacy of zoledronic acid on the biologic incorporation of cementless hip prosthesis in postmenopausal female patients.The study population consists of postmenopausal female patients scheduled for total hip replacement because of degenerative hip osteoarthritis. The patients will receive either a single dose of 5 mg zoledronic acid or placebo intravenously after surgery before hospital discharge. The patients will be followed-up for 1 year. Zoledronic acid therapy has been shown to promote bone ingrowth into porous implants in pre-clinical models. The investigators hypothesis is that zoledronic acid, given as a single intravenous infusion after hip replacement surgery, enhances bone ingrowth into porous surface of cementless hip prostheses. As a primary outcome, the therapy is expected to reduce periprosthetic bone loss measured by DXA. Enhancement of bone ingrowth is expected to increase primary stability of the hip prosthesis and this effect can be detected with high-precision three-dimensional RSA imaging modality and in a faster functional recovery of the patients.

DETAILED DESCRIPTION:
All the patients enrolled in the study will receive the standard of care with respect to surgical prosthetic replacement of the diseased hip. The patients will receive a custom-modified (RSA marked) hydroxyapatite-coated prosthesis with ceramic-on-ceramic bearing surfaces (SYMAX-TRIDENT, Stryker). The prosthesis modification provided by the manufacturer has a CE mark. The patients in the active-treatment group will receive a single 5 mg dose of zoledronic acid intravenously just prior to release from the hospital (about 5th day post-surgery) as an adjunct therapy. The control group will receive a placebo (saline) infusion. The active and placebo infusion vials will be provided by Norvartis Pharmaceutical. After surgery, before the administration of zoledronic acid or placebo, each patient will be re-screened for the level of serum calcium. In the case of postoperative hypocalcemia, the infusion will be postponed for a minimum of 3-4 weeks and the infusion will be given after the repeated measurements of serum calcium. All patients will receive calcium and D-vitamin supplementation throughout the study period. Efficacy will be assessed on the basis of clinical, radiographic (RSA, DXA, Spiral CT, conventional radiography) and laboratory criteria. The clinical benefit of zoledronic acid therapy is defined in terms of faster functional recovery, which will be analyzed in two ways: (1) the functional outcome (muscle strength, gait analysis and pedometry) will be repeatedly evaluated before and after surgery, and (2) the subjective outcome of the procedure as well as the general health assessment will be determined at each follow-up visits using standardized outcome measures. The primary objective of this study is to test whether a single infusion of zoledronic acid reduces periprosthetic bone loss measured by DXA at 12 months. Statistical significance of differences in periprosthetic bone mineral density between active-treatment and placebo groups will be analyzed using repeated analysis of variance.

ELIGIBILITY:
Inclusion Criteria:

* Degenerative hip osteoarthritis as the indication for hip replacement
* Postmenopausal female patient
* Age of at least 20 years
* Signed Informed Consent

Exclusion Criteria:

* Evidence of secondary osteoporosis
* Clinical or laboratory evidence of hepatic or renal disease
* Disorders of parathyroid function, or D-vitamin metabolism
* History of malignancy, radiotherapy, or chemotherapy for malignancy (except for basal cell carcinoma of the skin) within the past 5 years
* No metastatic cancer or cancer diagnosed less than 2 years ago where treatment is still ongoing
* Administration for more than 7 days of drugs, which may interfere with bone metabolism:

  * cumulative dose of 500 mg of prednisone or equivalent within the last 6 months
  * calcitonin within the last 6 months
  * bisphosphonates for 30 days or more within the last 12 months
  * bone therapeutic doses of fluoride for 30 days or more within the last 24 months
* Rheumatoid arthritis or any other inflammatory arthritis
* History of osteogenesis imperfecta, multiple myeloma, or Paget's disease
* Active primary hyperparathyroidism
* History of uveitis, iritis, or chronic conjunctivitis
* History of retinopathy or nephropathy, especially in the presence of uncontrollable IDDM (Hb1AC > 10%)
* AST or ALT > 2X the upper limit of normal
* ALP > 1.5X the upper limit of normal
* Serum creatine > 2 mg/dl
* Creatine clearance < 40 ml/min
* Serum calcium > 11.0 mg/dL and < 8mg/dL
* Serum 25(OH)D < 15 ng/ml
* In subjects with HIV must have a plasma HIV-1 RNA level of < 5000, a CD4+ count of > 100 cells/mm3m and be receiving stable ART for a minimum of 12 weeks prior study entry, with no plan at study entry to significantly alter ART
* Allergy to zoledronic acid
* Severe dental problems or current dental infections or with recent or impending dental surgery within three months of dosing

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-05; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to test whether a single infusion of zoledronic acid reduces periprosthetic bone loss measured by DXA. | 12 months

SECONDARY OUTCOMES:
RSA outcome, functional recovery and metabolic treatment response | 12 months
  * to demonstrate that the treatment can enhance biologic incorporation of cementless hip prostheses as shown by reduced prosthetic migration measured by RSA (radiostereometry)
  * to demonstrate that enhanced incorporation of the hip prostheses following the therapy lead to faster functional recovery and better subjective outcome of the procedure.
  * to demonstrate that the treatment suppresses biochemical markers of bone resorption.

CONTACTS AND LOCATIONS:
Overall Officials: Hannu T Aro, MD, PhD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland

REFERENCES:
- [Background] Makinen TJ, Alm JJ, Laine H, Svedstrom E, Aro HT. The incidence of osteopenia and osteoporosis in women with hip osteoarthritis scheduled for cementless total joint replacement. Bone. 2007 Apr;40(4):1041-7. doi: 10.1016/j.bone.2006.11.013. Epub 2007 Jan 17. PMID 17239668
- [Background] Makinen TJ, Koort JK, Mattila KT, Aro HT. Precision measurements of the RSA method using a phantom model of hip prosthesis. J Biomech. 2004 Apr;37(4):487-93. doi: 10.1016/j.jbiomech.2003.09.004. PMID 14996560
- [Background] Alm JJ, Makinen TJ, Lankinen P, Moritz N, Vahlberg T, Aro HT. Female patients with low systemic BMD are prone to bone loss in Gruen zone 7 after cementless total hip arthroplasty. Acta Orthop. 2009 Oct;80(5):531-7. doi: 10.3109/17453670903316801. PMID 19916684
- See also: Orthopaedic Research Unit — http://www.orthopaedics.utu.fi